CLINICAL TRIAL: NCT05831410
Title: The Role of Licensing in Early Care and Education (TRLECE): Survey of State and Territory Child Care and Early Education Licensing Administrators
Brief Title: The Role of Licensing in Early Care and Education: Licensing Administrators
Acronym: TRLECE:LA
Status: Completed | Type: Observational
Sponsor: Child Trends (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); ICF International, Inc. (Unknown)
Responsible Party: Principal Investigator, Kelly Maxwell, Senior Scholar, Early Childhood Research, Child Trends
Other Study IDs: 17187001; 233201500034I-75P00119F37007 (Other Grant/Funding Number: OPRE, ACF, US Dept. Health and Human Services (HHSP))
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Licensing Administrator Perceptions of the Licensing System
Keywords: Child care and early education; Child care licensing; Early care and education programs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Child Trends, funded by the Office of Planning, Research, and Evaluation (OPRE), Administration for Children and Families (ACF) in the U.S. Department of Health and Human Services (HHS) will collect descriptive information for The Role of Licensing in Early Care and Education (TRLECE): Licensing Administrators project. The goal of this information collection is to deepen the field's understanding of child care and early education licensing systems, which play a critical role in supporting positive outcomes for providers, families, and children. The investigators will conduct one round of survey data collection with all state and territory child care and early education licensing administrators.

DETAILED DESCRIPTION:
This study aims to advance understanding of the landscape of child care and early education licensing systems. State/territory child care and early education licensing agencies establish and monitor regulations that child care programs serving young children must meet to operate legally. These regulations and monitoring practices play a large role in the operations of child care programs but have received relatively little research attention. The field has limited information about features of state/territory licensing units and the characteristics and perceptions of licensing administrators. TRLECE: Licensing Administrators findings can inform licensing policies and practices in the child care and early education field, guidance and technical assistance to state leaders, and future research.

For this descriptive study, the investigators will conduct a survey of child care licensing administrators. This survey is designed to collect information about licensing administrator demographics, licensing agency structure and staff supports, ideas about the factors that influence decision-making, perceptions of strengths and challenges of the licensing system, and ideas to improve the licensing system. The investigators will invite the licensing administrator from each state and territory (n = 56) to participate.

ELIGIBILITY:
Inclusion Criteria:

* Child care licensing administrators in all U.S. states, territories, and the District of Columbia (DC)

Exclusion Criteria:

* Individuals who are not child care licensing administrators in all U.S. states, territories, and the District of Columbia (DC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Child care licensing administrators
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Child care licensing administrator survey | one time
  Survey developed by the study team to gather information about licensing processes and policies as well as administrators' characteristics, perceptions of their role, and ideas for improving licensing

CONTACTS AND LOCATIONS:
Overall Officials: Kelly L Maxwell, PhD, Principal Investigator — Child Trends
Locations (1):
- Child Trends Headquarters, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared. Information collected from Part 1 of this survey focuses on state/territory licensing system (e.g., structure, function, and regulations) and will be reported publicly and shared with the Child & Family Data Archive (CFData). Part 2 of the survey focuses on administrator perceptions and ideas. We anticipate that these data will be shared via a restricted use data set with the CFData Archive.
Time Frame: The team anticipates submitting IPD and supporting information to Child and Family Data Archive (CFData) roughly 6 months after the end of data collection. Data will be available after being reviewed by CFData. No end date on the availability of the data.
Access Criteria: Some data from the child care licensing administrator survey will be archived as public-use data with CFData and accessible on their website. Some data will be available as restricted-use only, following guidelines from CFData. Data will be shared with researchers for analyses related to child care licensing systems and experiences and perceptions of licensing administrators.